CLINICAL TRIAL: NCT03062072
Title: Emergence of Chemotherapy Related Hyperglycemia in nOn-diabetic Patients (ECHO)
Brief Title: Emergence of Chemotherapy Related Hyperglycemia in nOn-diabetic Patients
Acronym: ECHO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Eun Kyung Lee, Principal Investigator, National Cancer Center, Korea
Other Study IDs: ECHO; NCC2015-0040 (Other: NCC Korea)
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Cancer; Colon Cancer; Breast Cancer; Malignant Lymphoma
Keywords: normoglycemia; cancer; chemotherapy; Hyperglycemia Drug Induced
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Breast Neoplasms; Lymphoma | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, buffy coat
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chemotherapy — Chemotherapy containing glucocorticoid as anti-emetics or anti-cancer agent except for targeted agents
  Other Names: cytotoxic chemotherapeutic agents

SUMMARY:
To assess chemotherapy related hyperglycemia in non-diabetic patients, the investigators will assess the incidence of hyperglycemia and analyze co-medications and risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancers (colorectal, breast) who treated with curative intents and ones with malignant lymphoma who are expected to achieve complete remission with chemotherapy (mainly, CHOP regimen)
* Patients without history of diabetes mellitus
* Normal glucose tolerance, as defined in the protocol

Exclusion Criteria:

* Patients with diabetes mellitus or hyperglycemia, as defined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with advanced cancers (colorectal, breast) who treated with curative intents, and ones with malignant lymphoma who are expected to achieve complete remission with chemotherapy (mainly, CHOP regimen)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of type 2 diabetes mellitus | during chemotherapy (about 1 year)
  Percentage of patients who progressed to type 2 diabetes

SECONDARY OUTCOMES:
Change in HbA1c | during chemotherapy (about 1 year)
Change in glycated albumin | during chemotherapy (about 1 year)
Recurrence free survival (RFS) | from the Date of enrollment to the date of disease recurrence or date of any cause assessed upto 100 months

CONTACTS AND LOCATIONS:
Overall Officials: Eun Kyung Lee, Principal Investigator — National Cancer Center, Korea
Locations (2):
- South Korea (2):
  - National Cancer Center, Korea, Goyang
  - Seoul National University Boramae Medical Center, Seoul

REFERENCES:
- [Derived] Lee EK, Koo B, Hwangbo Y, Lee YJ, Baek JY, Cha YJ, Kim SY, Sim SH, Lee KS, Park IH, Lee H, Joo J, Go S, Heo SC, Moon MK. Incidence and disease course of new-onset diabetes mellitus in breast and colorectal cancer patients undergoing chemotherapy: A prospective multicenter cohort study. Diabetes Res Clin Pract. 2021 Apr;174:108751. doi: 10.1016/j.diabres.2021.108751. Epub 2021 Mar 17. PMID 33722701